CLINICAL TRIAL: NCT00291603
Title: Short-Term Effects of the FX-Class of Haemodialyser on Quality of Life and Inflammatory Markers in Stable Dialysis Patients
Brief Title: Short Term Effects of FX Dialysers on QOL and Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Charles Gairdner Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-192
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Kidney Failure, Chronic
Keywords: dialysis; Renal Dialysis; inflammation; quality of life; End Stage Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FX-class of dialyser

SUMMARY:
Background:

The new hollow fibre FX-class of dialysers (Fresenius Medical Care, Bad Homburg, Germany) features a number of technological improvements that may benefit the patient. This includes the use of the advanced high-flux polysulfone membrane, Helixone®, which has an extremely high endotoxin retaining capability. Theoretically leading to reduced systemic inflammation in the patient, which is an important factor for morbidity and mortality with dialysis.

The dialysis membrane is the first to be manufactured using membrane-spinning procedures (nano-controlled spinning technology) that enables the membrane to be modulated at the nano-scale level. The resultant membrane is able to extremely efficiently remove middle molecules, along with minimal loss of albumin.

These features may lead to improved patient outcomes, including reduced systemic inflammation and improved quality of life.

Aims:

1. To assess the short-term effects of the FX-class Dialyser on quality of life in stable haemodialysis patients
2. To assess the short-term effects of the FX-class Dialyser on inflammatory markers in stable haemodialysis patients.

DETAILED DESCRIPTION:
Methods Patient selection All patients in the Joondalup Health Campus satellite dialysis unit will be invited to participate in this study.

Inclusion criteria -

1. Age >18years
2. Able to provide informed consent
3. On haemodialysis for 3 months

Exclusion criteria -

1. Active inflammatory, infective or neoplastic process within the last 1 month
2. Active major psychiatric condition
3. Currently on haemodiafiltration as haemodialysis modality

Design This study will involve an unblinded, cross-over design, with patients being randomised upon entry into one of 2 groups. The 2 groups will be - 1. HF80 dialyser (this is the best of the currently used dialysers and therefore no participant will require a reduction in their dialysis during this trial); and 2. FX dialyser. Patients will have baseline tests performed prior to intervention and then repeated after 3 months. At 3 months, patients will then cross-over into the other group and tests repeated after a further 6 months.

Due to the nature of the intervention, blinding will not be practical. The cross-over design will allow maximum power for this fixed and relatively small dialysis population (~50 patients).

Independent variables -

1. Dialysis prescription on enrolment

   a. Including dialyser type (biocompatibility)
2. Adequacy of dialysis

   1. Urea reduction ratio
   2. Kt/V
3. Anaemia

   1. Including iron studies
   2. Including erythropoietin usage
4. Calcium phosphate balance

   a. Including Parathyroid hormone levels
5. Serum albumin

Outcome markers -

1. Quality of Life (i) KD-QOL - this is a standardised quality of life questionnaire designed and validated for dialysis patients, that will be readily comparable to other studies.

   (ii) Feeling thermometer
2. Inflammatory markers (i) High sensitivity c-reactive protein (ii) IL-6 (iii) White cell count.

Statistical analysis:

Quality of life measures and inflammatory markers will be analysed using paired t-test after normality demonstrated. Simple and multiple linear regression analysis will then be performed to examine associations between independent variables with changes in the outcome variables. STATA 8.2 will be used to assist with the analysis

ELIGIBILITY:
Inclusion Criteria:

1. Age >18years
2. Able to provide informed consent
3. On haemodialysis for 3 months

Exclusion Criteria:

1. Active inflammatory, infective or neoplastic process within the last 1 month
2. Active major psychiatric condition
3. Currently on haemodiafiltration as haemodialysis modality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-02; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
KD-QOL
Feeling Thermometer

SECONDARY OUTCOMES:
IL-6
TNF-alpha
hs-CRP
white cell count

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Boudville, MD, Principal Investigator — The University of Western Australia
Locations (1):
- Joondalup Health Campus Satellite Dialysis Unit, Perth, Western Australia, Australia